CLINICAL TRIAL: NCT04818450
Title: Impact of Gabapentin on Slow Wave Sleep in Adult Critically Ill Patient.
Acronym: GASWAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MURA2021/170
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Sleep Deprivation; Critically Ill
Keywords: gabapentin; sleep deprivation; critically ill patients; slow-wave sleep
MeSH Terms: conditions — Sleep Deprivation; Critical Illness | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): Start gabapentin 100 mg at 9.00 PM on the second night of ICU admission and titrate gabapentin dose as needed. Maximum gabapentin dose in this study is 300 mg/day.
  Interventions: Drug: Gabapentin
- Standard care (No Intervention): Not receiving gabapentin.

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 100-300 mg is given to the intervention group
  Other Names: Gabapentin group
  Arms: Gabapentin

SUMMARY:
The investigators proposed that gabapentin will increase slow-wave sleep in adult critically ill patients. Increasing slow-wave sleep will improve the patients' outcomes (shortening ICU length of stay, improving ventilator free days, increasing delirium free days) in critically ill patients, a university hospital, Thailand.

DETAILED DESCRIPTION:
Up to 61% of critically ill patients have sleep deprivation in ICU. Sleep deprivation can cause delirium and lead to prolonged ICU length of stay and mechanical ventilator days. However, pharmacologic interventions to improve sleep quality and prevent sleep deprivation are poorly tested for efficacy and safety in ICU patients. There were reports of gabapentin increasing slow-wave sleep in healthy populations and insomnia patients with insignificant adverse events. Therefore, gabapentin might increase slow-wave sleep resulting in improving clinical outcomes in adult critically ill patients. The objectives of the study were to evaluate the efficacy, especially on slow-wave sleep, and safety of gabapentin in adult critically ill patients admitted to ICUs at Ramathibodi Hospital, a university hospital, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Patients admitted to ICU not more than 24 hours at the time of randomization

Exclusion Criteria:

* Patients admitted to ICU less than 72 hours
* Patients receiving gabapentin within 14 days prior to randomization
* Patients receiving restorative drug (trazodone, mirtazapine, olanzapine, agomelatine, and pregabalin) within 7 days prior to randomization
* Patients having contraindications to gabapentin
* Patients receiving high dose vasopressors more than 1 hour during ICU admissions
* Patients presenting with severe respiratory failure (PF ratio < 100)
* Patients presenting with RASS < -2 at the time of randomization
* Patients having target RASS of <-2 during ICU admissions
* Terminal ill patients
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Slow-wave sleep | at least 3 consecutive days after randomization
  Slow-wave sleep period or deep sleep period

SECONDARY OUTCOMES:
All-cause hospital mortality | During hospital stay or death or a maximum of 90 days
  Rates of all-cause mortality during hospital stay
ICU free days | During ICU stay or death or a maximum of 28 days
  Days alive and not stay in ICU
Mechanical ventilator free days | During ICU stay or death or a maximum of 28 days
  Day alive and free of mechanical ventilator
Hospital free days | During hospital stay or death or a maximum of 90 days
  Days alive and not stay in hospital
Incidence of self-extubation | During ICU stay or death or a maximum of 28 days
  Number of patients who had self-extubation during ICU stay
Incidence of sleep deprivation | During ICU stay or death or a maximum of 28 days
  Times per patient-days of sleep deprivation during ICU stay
Delirium free day | During ICU stay or death or a maximum of 28 days
  Days alive and not having delirium

OTHER OUTCOMES:
IGF-1 | At day 0, 1, 3, and 5 after randomization
  IGF-1 level

CONTACTS AND LOCATIONS:
Overall Officials: Yuda Sutherasan, MD, Study Director — Ramathibodi hospital, Mahidol university; Kanyarat Susantitapong, B.Sc.(Pharm), Principal Investigator — Mahidol University; Pitchaya Dilokpattanamongkol, BCPS, BCCCP, BCP, Study Director — Mahidol University; Chuthamanee Suthisisang, Ph.D., Study Chair — Mahidol University; Viratch Tangsujaritvijit, Ph.D., Study Chair — Piyavate Hospital
Locations (1):
- Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Arttawejkul P, Reutrakul S, Muntham D, Chirakalwasan N. Effect of Nighttime Earplugs and Eye Masks on Sleep Quality in Intensive Care Unit Patients. Indian J Crit Care Med. 2020 Jan;24(1):6-10. doi: 10.5005/jp-journals-10071-23321. PMID 32148342
- [Result] Carrera-Hernandez L, Aizpitarte-Pejenaute E, Zugazagoitia-Ciarrusta N, Goni-Viguria R. Patients' perceptions of sleep in a Critical Care Unit. Enferm Intensiva (Engl Ed). 2018 Apr-Jun;29(2):53-63. doi: 10.1016/j.enfi.2018.01.002. Epub 2018 Mar 28. English, Spanish. PMID 29605589
- [Result] Foldvary-Schaefer N, De Leon Sanchez I, Karafa M, Mascha E, Dinner D, Morris HH. Gabapentin increases slow-wave sleep in normal adults. Epilepsia. 2002 Dec;43(12):1493-7. doi: 10.1046/j.1528-1157.2002.21002.x. PMID 12460250
- [Result] Liu GJ, Karim MR, Xu LL, Wang SL, Yang C, Ding L, Wang YF. Efficacy and Tolerability of Gabapentin in Adults with Sleep Disturbance in Medical Illness: A Systematic Review and Meta-analysis. Front Neurol. 2017 Jul 14;8:316. doi: 10.3389/fneur.2017.00316. eCollection 2017. PMID 28769860
- [Result] Rosenberg RP, Hull SG, Lankford DA, Mayleben DW, Seiden DJ, Furey SA, Jayawardena S, Roth T. A randomized, double-blind, single-dose, placebo-controlled, multicenter, polysomnographic study of gabapentin in transient insomnia induced by sleep phase advance. J Clin Sleep Med. 2014 Oct 15;10(10):1093-100. doi: 10.5664/jcsm.4108. PMID 25317090
- [Result] Lo HS, Yang CM, Lo HG, Lee CY, Ting H, Tzang BS. Treatment effects of gabapentin for primary insomnia. Clin Neuropharmacol. 2010 Mar-Apr;33(2):84-90. doi: 10.1097/WNF.0b013e3181cda242. PMID 20124884
- [Derived] Susantitapong K, Dilokpattanamongkol P, Sutherasan Y, Liamsombut S, Suthisisang C. Effects of gabapentin on slow-wave sleep period in critically ill adult patients: A randomized controlled trial. Clin Transl Sci. 2024 May;17(5):e13815. doi: 10.1111/cts.13815. PMID 38803031